CLINICAL TRIAL: NCT01518686
Title: Normal Values for the Full Visual Field, Corrected for Age- and Reaction Time, Using Semi-automated Kinetic Testing on the Octopus 900 Perimeter
Brief Title: Age-related Normative Values for the Octopus 900 Perimeter
Acronym: Norm-Oct900
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Collaborators: Haag-Streit AG (Industry)
Responsible Party: Principal Investigator, Ulrich Schiefer, Prof. Dr. med Ulrich Schiefer, University Hospital Tuebingen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 217/2006 local review board
Record Dates: First submitted 2012-01-12; First posted 2012-01-26 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-12

CONDITIONS: Healthy
Keywords: Norm values; semi-automated kinetic perimetry; isopters; mathematical model; luminance; test-retest reliability; deviation; age dependance; different age groups; Healthy subjects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- one arm (No Intervention): observational study, no cohort, single group of different ages
  Interventions: Device: Octopus 900 perimeter (Haag Streit AG, Koeniz, Switzerland)

INTERVENTIONS:
Device: Octopus 900 perimeter (Haag Streit AG, Koeniz, Switzerland) — We used the following six combinations of Goldmann8,1 stimulus size, stimulus luminance and angular velocity: V4e (64mm², 103', 320cd/m²) at 5°/s, III4e (4mm², 25.7', 320cd/m²) at 5°/s, I4e (0.25mm², 6.45', 320cd/m²) at 2°/s (for the assessment of the blind spot), I3e (0.25mm², 6.45', 100cd/m²) at 5°/s, I2e (0.25mm², 6.45', 32cd/m²) at 3°/s, I1e (0.25mm², 6.45', 10cd/m²) at 3°/s, I1a (0.25mm², 6.45', 4cd/m²) at 2°/s .
  The peripheral five isopters, consisting of 24 vectors (every 15° meridian), were presented in random order, while the innermost isopter (I1a) consisted of 12 vectors (every 30° meridian)

SUMMARY:
The purpose of this study is to determine normal values of the visual field (VF), corrected for age- and reaction time (RT) using the Octopus 900 perimeter and semi-automated kinetic perimetry (SKP).

ELIGIBILITY:
Inclusion Criteria:

* maximum spherical ametropia ± 6 Diopters (D)
* maximum cylindrical ametropia ± 2 D
* distant visual acuity ≥ 1.0 logMAR [20/20] for subjects up to 60 years, ≥ 0.8 logMAR [20/25] for subjects from 61-70 years, ≥ 0.63 logMAR [20/30] for subjects older than 70 years
* isocoria, pupil diameter > 3mm
* intraocular pressure (air pulse tonometer) ≤ 21mmHg
* normal anterior segments
* ocular fundus: normal appearance of the cup to disc ratio (CDR) ≤ 0.5, interocular difference of CDR < 0.3
* normal macular region, vessels, and peripheral retinal examination (with undilated pupils).

Exclusion Criteria:

* amblyopia
* strabismus
* ocular motility disorder
* diseases of the retina
* glaucoma, glaucoma suspect
* macular degeneration
* IOP > 21 mmHg
* abnormal color vision test (ISPP - Ishihara and Standard Pseudoisochromatic Plates = SPP)
* history or findings of other neuro-ophthalmological disease
* relevant opacities of the central refractive media (cornea, lens, vitreous body)
* use of miotic drugs
* intraocular surgery (except uncomplicated cataract surgery, more than three months previous to testing)
* kerato-refractive surgery (LASIK)
* drugs influencing reaction time
* drugs indicating severe general diseases (anti-diabetic pharmaceuticals and anti-hypertensive medication were allowed for subjects older than 70 years)
* mental diseases (for example psychosis)
* pregnancy, nursing
* acute infections
* heavy smoking (>10 cigarettes /day)
* alcohol abuse
* diabetic retinopathy
* coronary heart disease
* stroke
* migraine
* Raynaud's syndrome
* suspected lack of compliance

Ages: 11 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2006-06; Primary Completion 2008-03 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Measurement of the full Visual Field using semi-automated kinetic perimetry. | one day
  additional a subgroup of 14 participants were tested at 3 separate sessions within 4 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich Schiefer, Prof. Dr. med., Principal Investigator — Centre for Ophthalmology / Institute for Ophthalmic Research, University of Tübingen, Germany
Locations (1):
- Centre for Ophthalmology / Institute for Ophthalmic Research, University of Tübingen, Tübingen, Baden-Wurttemberg, Germany